CLINICAL TRIAL: NCT03207698
Title: Evaluation of Adjunctive Effect of 1% Metformin To Platelet Rich Fibrin For Mandibular Class II Furcation Defects: A Randomized Controlled Clinical Trial
Brief Title: PRF+1% MF for Class II Mandibular Furcation Defects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and Head, Dept of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014KD
Record Dates: First submitted 2017-07-01; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Furcation Defects
MeSH Terms: conditions — Furcation Defects | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Scaling and Root Planing (SRP) with Open flap debridement (OFD) alone for treating furcation defect
  Interventions: Procedure: Open flap debridement (OFD)
- Group 2 (Active Comparator): SRP with Open flap debridement (OFD) with Platelet rich fibrin (PRF) for treating furcation defect
  Interventions: Procedure: OFD with Platelet rich fibrin (PRF)
- Group 3 (Active Comparator): SRP with Open flap debridement (OFD) with Platelet rich fibrin (PRF)+1% Metformin for treating furcation defect
  Interventions: Procedure: OFD with Platelet rich fibrin (PRF)+1% Metformin (Drug) in gel form

INTERVENTIONS:
Procedure: Open flap debridement (OFD) — Open flap debridement (OFD) alone
  Arms: Group 1
Procedure: OFD with Platelet rich fibrin (PRF) — Open flap debridement (OFD) with Platelet rich fibrin (PRF) placement
  Arms: Group 2
Procedure: OFD with Platelet rich fibrin (PRF)+1% Metformin (Drug) in gel form — Open flap debridement (OFD) with Platelet rich fibrin (PRF)+1.2% Atorvastatin gel placement
  Arms: Group 3

SUMMARY:
The aim of the present trial is to evaluate the efficacy of PRF with 1% MF in treatment of mandibular class II furcation defects and its comparison to PRF and access therapy alone.

DETAILED DESCRIPTION:
Background: For improving efﬁcacy and outcomes of regenerative therapy for furcation defects, various materials has been investigated in addition to access therapy. Platelet-rich fibrin (PRF) having concentrated growth factors and cytokines and Metformin (MF), an efficacious member of biguanide group are known to enhance periodontal regeneration. The aim of the present trial is to evaluate the efficacy of PRF with 1% MF in treatment of mandibular class II furcation defects and its comparison to PRF and access therapy alone.

Methods: This randomized trial was conducted on 75 patients with mandibular class II furcation defects. Defects were surgically treated with either access therapy alone (Group 1), access therapy+PRF (Group 2), and access therapy+ PRF+1% MF (Group 3). Clinical parameters like probing depth (PD), relative clinical attachment level {vertical (RVCAL) and horizontal (RHCAL)}, modified sulcus bleeding index (mSBI) and site specific plaque index (PI) were evaluated at baseline and 9 months post-operatively. Radiological assessment of bone defect fill was done at baseline and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Buccal degree II furcation defects in endodontically vital, asymptomatic mandibular first and second molars with a radiolucency in the furcation area on an intraoral periapical radiograph with probing depth (PD) ≥ 5mm and horizontal ≥ PD 3mm after phase I therapy i.e, scaling and root planing (SRP);
* No history of antibiotic or periodontal therapy in the preceding 6 months.

Exclusion Criteria:

Aggressive periodontitis patients

* Systemic conditions known to affect the periodontal status;
* Medications known to affect the outcomes of periodontal therapy;
* Hematological disorders and insufficient platelet count (<100,000/mm3);
* Pregnancy/lactation;
* Smoking and tobacco use in any form
* Immunocompromised individuals;
* Those having unacceptable oral hygiene (plaque index [PI] >1.5).
* Teeth with furcation involvement, non-vital teeth, and carious teeth indicated for restorations and mobility of at least grade II were also excluded.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Radiographic bone fill assessed in percentage | baseline to 9 months
  assessed in percentage

SECONDARY OUTCOMES:
probing depth measured in mm | baseline to 9 months
  measured in mm
Relative vertical attachment level measured in mm | baseline to 9 months
  measured in mm
Relative horizontal attachment level measured in mm | baseline to 9 months
  measured in mm
modified sulcus bleeding index | baseline to 9 months
  0-3 scale
plaque index | baseline to 9 months
  0-3 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India